CLINICAL TRIAL: NCT05547191
Title: An Open, Single-arm, Multicentre and Interventional Investigation to Evaluate the Debriding Effect of ChloraSolv® on Pressure Ulcers in Need of Debridement
Brief Title: Evaluate Efficacy and Safety of ChloraSolv When Treating Pressure Ulcers in Need of Debridement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: RLS Global in bankruptcy
Sponsor: RLS Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PN-00041; 320237 (Registry Identifier: IRAS Integrated Research Application System)
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-09

CONDITIONS: Pressure Ulcer
Keywords: Pressure ulcer; Debridement; ChloraSolv
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational device (Experimental): ChloraSolv
  Interventions: Device: ChloraSolv

INTERVENTIONS:
Device: ChloraSolv — Debridement with ChloraSolv until the wound is visually assessed as clean.

SUMMARY:
This is an open, single-arm, multicentre and interventional investigation to evaluate the debriding effect of ChloraSolv when used on pressure ulcers in need of debridement. Approximately 54 subjects will be enrolled to have 47 evaluable subjects (calculated dropout range 15%).

ChloraSolv will be applied 1-2 times per week for 12 weeks or until the wound is deemed clean, whichever occurs first i.e. End of Treatment. A Follow-up visit for wound status evaluation will be performed 6 weeks from End of Treatment. Total time in investigation will be maximum 12+6 weeks.

Subjects will attend a baseline visit to assess eligibility and collect demographic and baseline data and initiate treatment. Photographs of the wound pre and post debridement will be taken at baseline, every week during the treatment period, at End of Treatment and at the Follow-up visit. Photographs will be used to calculate (by PictZar digital planimetry system) the area of devitalized tissue in the wound as well as wound size and calculation of volume.

Wound depth and undermining will be estimated by the investigator at all investigational visits.

A treatment diary will be used in-between the weekly investigational visits to collect any further treatments. The treatment diary will also be filled-in during the follow-up period of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Pressure ulcer in need of debridement
2. Male or female, 18 years of age and above
3. Able to read and understand the Patient Informed Consent and to provide written informed consent. If written consent is not possible due to the condition of the patient, one impartial witness shall sign and date the informed consent.

Exclusion Criteria:

1. Known allergy/hypersensitivity to any of the components of ChloraSolv
2. Pregnancy or breastfeeding
3. Subjects included in other ongoing clinical investigations which could interfere with this investigation, as judged by the investigator
4. Subjects not suitable for the investigation according to the investigator's judgment or other significant medical conditions that the investigator determines could interfere with compliance or investigation assessments
5. Wound requiring more than two (2) ChloraSolv syringes for one treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Incidence of subjects with a clean wound bed, not in need of further debridement at End of Treatment, as assessed by investigator | 1-12 weeks
  When the investigator judge that the wound is clean, primary endpoint is reached

SECONDARY OUTCOMES:
Incidence of subjects with a clean wound bed at End of Treatment, as assessed by planimetry | 1-12 weeks
  When the investigator judges that the wound is clean and this is confirmed by planimetry
Relative change in devitalized tissue at End of Treatment and Follow-up, compared to Baseline, assessed by planimetry | 1-18 weeks
  Changes in devitalized tissue, measured by planimetry
Relative change in wound area at End of Treatment and Follow-up, compared to Baseline and End of Treatment, assessed by planimetry | 1-18 weeks
  Changes in wound area, measured by planimetry
Relative change in volume at End of Treatment and Follow-up, compared to Baseline and End of Treatment, assessed by planimetry | 1-18 weeks
  Changes in volume, measured by planimetry
Relative change in wound depth and undermining at End of Treatment and Follow-up, compared to Baseline, assessed by investigator by using a sterile cotton-tipped applicator | 1-18 weeks
  Changes in wound depth (mm) and undermining (mm) will be measured by site personnel using a sterile cotton-tipped applicator and read against a wound ruler.
Pain during treatment compared to baseline using a Visual Analogue Scale | 1-12 weeks
  Changes in pain during treatment from baseline to End of Treatment. Minimum value=0 (No pain), Maximum value=100 (Worst imaginable pain)
Wound status i.e. clinical signs of infection at all visits | 1-18 weeks
  Clinical signs of infection will be documented by ticking off a list with five alternatives/symptoms (redness, heat, edema, pain and odour).Three or more symptoms will be assessed as the subject having clinical signs of infection.
Treatment period duration with ChloraSolv | 1-12 weeks
  Number of weeks that ChloraSolv was used
Number of treatments with ChloraSolv from Baseline until End of Treatment | 1-12 weeks
  Number of treatments with ChloraSolv until end of treatment
Incidence of subjects with complete wound healing during the investigation period | 1-18 weeks
  Number of patients receiving a healed wound
Incidence of subjects needing sharp debridement during the investigation period and compared to before start of the investigation | 0-18 weeks
  Usage of sharp (scalpel or knife) debridement during the investigation period
Answers from overall evaluation by site personnel | Through study completion, an average of 1 year
  A questionnaire consisting of 5 questions (evaluating the handling/usage of the investigational device) will be filled in by site personnel at end of investigation. There will be four alternatives; Very easy/Easy/Difficult/Very difficult
Answers from overall evaluation by subjects | 1-12 weeks
  The subjects will be asked to answer four questions (overall experience with the investigational device) at end of treatment. There will be four alternatives; Very good/Good/Bad/Very Bad

OTHER OUTCOMES:
Frequency, severity, device relationship and outcome of all adverse events | 0-18 weeks
  Collection of adverse events to evaluate safety

CONTACTS AND LOCATIONS:
Locations (6):
- Kirurgkliniken, Ålands hälso- och sjukvård, Mariehamn, Åland, Aland Islands
- Dept of Orthopaedic Surgery, Mölndal, Sweden
- United Kingdom (4):
  - Buckinghamshire Healthcare NHS Trust, Aylesbury, England
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool, England
  - East London NHS Foundation Trust, Newham, England
  - Greater Glasgow Health Board, Glasgow, Scotland